CLINICAL TRIAL: NCT05791279
Title: The Use of Electrocardiography-based Estimation of Heart Age to Improve Blood Pressure in a Primary Care Setting - a Pilot Study
Brief Title: Electrocardiography-based Estimation of Heart Age to Improve Blood Pressure - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Lund University (Other); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Kronoberg_HA
Record Dates: First submitted 2023-02-20; First posted 2023-03-30 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): The participants in the intervention group will receive information about their ECG-based Heart-Age and the Heart Age. The estimated Heart Age and Heart Age Gap will be presented in writing to the participants in the experimental arm within 2 weeks after the baseline visit. The presentation will include a brief and easy-to-understand description on how the Heart Age has been estimated. In addition, patients will receive information about general advice on how to improve blood pressure levels and reduce the risk of future cardiovascular disease by adopting a healthy lifestyle and adhering to the prescribed medication. This information will be the same for participants in the two study arms, and is based on recommendations from the European Society of Cardiology.
  For patients in the intervention group the ordinary primary care physicians will also be informed about the ECG-based Heart-Age.
  Interventions: Other: Heart age
- Control arm (No Intervention): The control group will receive standard care according to routine care at the individual primary health care center, and receive the same general advice, on how to improve blood pressure levels and/or to reduce risks of future cardiovascular disease, as the participants in the intervention group.

INTERVENTIONS:
Other: Heart age — information about their ECG-based Heart-Age and the Heart Age gap, i.e. the difference between chronological and ECG-based Heart Age.
  Arms: Interventional arm

SUMMARY:
Successfully communicating cardiovascular risk to patients is essential for achieving compliance to medication and lifestyle changes. An intuitive way to translate cardiovascular risk is to present a Heart Age; an ECG-based age-estimation from ECG changes which can be contrasted to a patient's chronological age. In this pilot study, the feasibility of a randomized controlled study (RCT) in which hypertensive patients in primary care will receive information about their ECG-based Heart Age in addition to standard care, or standard care alone, will be assessed, in preparation for a larger RCT.

DETAILED DESCRIPTION:
Cardiovascular disease processes begin early and progress silently for many years. Fortunately, several risk-factors are modifiable, and cardiovascular risk can therefore be reduced for example by smoking cessation, dietary changes, increased physical activity in sedentary people and adherence to pharmacological risk factor reduction. To accomplish this, the patient must understand that he or she is at risk. One way to do this could be to present the risk as a "Heart Age", which can be contrasted to the patient's chronological age. In a previous study, an accurate Heart Age could be obtained using conventional, 10-second ECG recordings. The ECG analysis included conventional and basic ECG measurements such as heart rate and waveform amplitudes and durations, but also combinations of advanced ECG measures from 12-lead-ECG-derived vectorcardiography and waveform complexity.

However, it is not known whether the use of Heart Age can improve outcomes if applied in clinical care. To address this issue, a study in which patients, in addition to standard care, are randomized to either being presented with their Heart Age or not should be performed. In order to check the feasibility of such a randomized controlled study (RCT), a pilot study is necessary.

This study will evaluate the feasibility of randomizing patients with hypertension to either being presented with their Heart Age or not, in addition to standard care, by describing the recruitment dropout rate, the quality of the recorded ECG and the tolerability of the intervention (participant experience).

At the baseline visit a standardized resting blood pressure, height, weight and waist circumference will be measured. Baseline characteristics (age, sex, hypercholesterolemia, diabetes, ischemic heart disease, cerebrovascular disease, renal failure, heart failure, medications) will be recorded from the patient records. Unless a recent (<1 month) ECG is available, a new resting ECG recording will be performed, and blood sampling will be done (total cholesterol, high-density lipoprotein [HDL], low-density lipoprotein [LDL] mmol/l, triglyceride mmol/mol, Hba1c (IFCC) mmol/mL, P-Creatinine (µmol/L). The participant will also receive a questionnaire for background information and information about tobacco and alcohol use, level of physical activity, dietary habits, medication adherence, quality of life and self-estimated health including estimating one's own risk of cardiovascular morbidity.

ECG-based Heart Age will be estimated for all participants but presented only to patients in the intervention arm. A follow-up visit will be performed 6 months after the baseline visit. At follow-up, the same measurements including the same questionnaires will be obtained. Participants in the intervention arm will also receive a questionnaire on their experience of receiving information about their Heart Age (tolerability).

ELIGIBILITY:
Eligibility: Patients with hypertension and systolic blood pressure >140 mm Hg (measured during the inclusion period by doctor or nurse at the primary health care center)

Inclusion Criteria:

* Informed consent
* Diagnosed hypertension (International classification of disease (ICD-10), I10.9)
* 40 - 75 years

Exclusion Criteria:

* ECG findings that are incompatible with or may significantly distort the Heart Age estimation (left/right bundle branch block, atrial fibrillation/flutter, tachycardia (≥100/min), abundant ventricular ectopic beats, misplaced ECG electrodes, missing leads, excessive signal noise/baseline)
* Short life expectancy (<1 year)
* Pregnancy, known secondary hypertension
* Predicted inability to give informed consent due to either language difficulties, cognitive impairment or other.
* Systolic blood pressure <120 mmHg at the baseline visit

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  Number of patients being recruited within the specified time frame
Dropout rate | 6 months
  Number of patients who do not complete follow-up
Quality | 6 months
  Number of Heart Age estimations with adequate ECG signal quality
Tolerability of the intervention | 6 months
  Tolerability of the intervention assessed through questionnaires.

SECONDARY OUTCOMES:
Blood pressure (systolic and diastolic) | 6 months
  Change in blood pressure
HbA1c | 6 months
  Change in HbA1c
Physical activity | 6 months
  Change in physical activity assessed through questionnaires.
Dietary habits | 6 months
  Change in dietary habits assessed through questionnaires.
Tobacco | 6 months
  Change in tobacco use assessed through questionnaires.
Alcohol | 6 months
  Change in alcohol use assessed through questionnaires.
Medication adherence | 6 months
  Change in medication adherence assessed through questionnaires.
Risk perception | 6 months
  Change in risk perception assessed through questionnaires.
Body-mass index (BMI) | 6 months
  Change in BMI
Heart Age | 6 months
  Change in Heart Age

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lindow, MD, PhD, Principal Investigator — Region Kronoberg, Sweden; Lund University, Lund, Sweden
Locations (2):
- Sweden (2):
  - Ryd Vardcentral, Ryd
  - Tingsryd Vardcentral, Tingsryd

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindow T, Palencia-Lamela I, Schlegel TT, Ugander M. Heart age estimated using explainable advanced electrocardiography. Sci Rep. 2022 Jun 14;12(1):9840. doi: 10.1038/s41598-022-13912-9. PMID 35701514